CLINICAL TRIAL: NCT00010101
Title: INI1 Mutation Analysis and Expression Profiling of Embryonal CNS Tumors
Brief Title: Genetic Study of Brain Tumors in Young Children
Status: Terminated | Type: Observational
Why Stopped: Poor accrual
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: James M. Boyett/PBTC Operations and Biostatistics Center Executive Director, Pediatric Brain Tumor Consortium
Other Study IDs: CDR0000068445; PBTC-N03
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Central Nervous System Tumor, Pediatric
Keywords: childhood choroid plexus tumor; untreated childhood supratentorial primitive neuroectodermal tumor; untreated childhood medulloblastoma; childhood atypical teratoid/rhabdoid tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Choroid Plexus Neoplasms; Rhabdoid Tumor

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Tumor samples
Oversight: Data Monitoring Committee: No

SUMMARY:
RATIONALE: Genetic studies may help in understanding the genetic processes involved in the development of some types of cancer.

PURPOSE: Genetic study to understand how genes may be involved in the development of brain tumors in young children.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the frequency and type of deletions and mutations of the INI1 gene in infants with embryonal central nervous system tumors.
* Compare the gene expression profiles in infants with atypical teratoid/rhabdoid tumors vs medulloblastoma or primitive neuroectodermal tumor.

OUTLINE: This is a multicenter study.

Tumor samples are analyzed by fluorescence in situ hybridization (FISH) for deletions of INI1 gene in chromosome band 22q11.2. Tumors without demonstration of deletions of INI1 gene by FISH are examined by polymerase chain reaction (PCR)-based microsatellite analysis for loss of heterozygosity using markers that map to 22q11.2.

DNA from tumor tissue is analyzed for mutations in the exons of the INI1 gene. Isolated matched normal DNA may be analyzed for identification of germline mutations. Parental DNA may be analyzed to identify inherited germline mutations of the INI1 gene.

The patient's physician may receive the results of the genetic testing. The results do not influence the type or duration of treatment.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 25 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary intracranial central nervous system tumor

  * Medulloblastoma
  * Primitive neuroectodermal tumor
  * Atypical teratoid/rhabdoid tumor
  * Choroid plexus carcinoma
* Potential enrollment on PBTC-001 therapeutic protocol

PATIENT CHARACTERISTICS:

Age:

* Under 3

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior steroids allowed

Radiotherapy:

* No prior radiotherapy

Surgery:

* Not specified

Other:

* No concurrent investigational agents

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Tissue samples from infants (< 3 years old) with histologically confirmed primary intracranial CNS medulloblastoma/PNET, atypical teratoid/rhabdoid tumor, or choroid plexus carcinoma and with no prior chemotherapy, radiotherapy, or treatment from any other investigational agent will be used for this research study. Patients who meet the eligibility criteria, are treated at a PBTC institution that has IRB approval of this study, and consent to the usage of stored tumor specimens for the study objectives constitute the study population.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2001-03; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Deletions and mutations of the INI1 gene in infants with AT/RT, medulloblastoma, PNET, or choroid plexus carcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Jaclyn A. Biegel, PhD, Study Chair — Children's Hospital of Philadelphia
Locations (4):
- United States (4):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Cancer Center, Houston, Texas

REFERENCES:
- [Result] Pomeroy SL, Tamayo P, Gaasenbeek M, Sturla LM, Angelo M, McLaughlin ME, Kim JY, Goumnerova LC, Black PM, Lau C, Allen JC, Zagzag D, Olson JM, Curran T, Wetmore C, Biegel JA, Poggio T, Mukherjee S, Rifkin R, Califano A, Stolovitzky G, Louis DN, Mesirov JP, Lander ES, Golub TR. Prediction of central nervous system embryonal tumour outcome based on gene expression. Nature. 2002 Jan 24;415(6870):436-42. doi: 10.1038/415436a. PMID 11807556